CLINICAL TRIAL: NCT00347932
Title: A Study to Evaluate the Clinical and Microbial Efficacy of 0.6% ISV-403 Compared to Vehicle in the Treatment of Bacterial Conjunctivitis.
Brief Title: A Study to Determine if 0.6% ISV-403 is Safe and Effective in the Treatment of Bacterial Conjunctivitis.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Bausch & Lomb Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 433; BOL-303224 (Registry Identifier: CAS)
Record Dates: First submitted 2006-06-30; First posted 2006-07-04 (Estimated); Results first posted 2009-08-13 (Estimated); Last update posted 2015-03-24 (Estimated); Status verified 2015-03

CONDITIONS: Acute Bacterial Conjunctivitis
MeSH Terms: interventions — besifloxacin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- ISV-403 (Experimental): 0.6% ISV-403 ophthalmic suspension
  Interventions: Drug: ISV-403
- Vehicle (Placebo Comparator): Vehicle of ISV-403 ophthalmic suspension
  Interventions: Drug: Vehicle

INTERVENTIONS:
Drug: ISV-403 — Subjects with bacterial conjunctivitis were randomized to receive 0.6% ISV-403 eye drops three times a day (TID) for 5 days.
  Other Names: besifloxacin; Besivance; BOL-303224
  Arms: ISV-403
Drug: Vehicle — Subjects with bacterial conjunctivitis were randomized to receive vehicle eye drops three times a day (TID) for 5 days.
  Arms: Vehicle

SUMMARY:
Evaluation of the clinical and microbial efficacy of 0.6% ISV-403, compared to vehicle in the treatment of bacterial conjunctivitis.

ELIGIBILITY:
Inclusion Criteria:

* Must have a diagnosis of acute bacterial conjunctivitis and exhibit purulent conjunctival discharge and redness in at least one eye.
* Females of childbearing potential must utilized reliable contraceptive methods and have a negative pregnancy test.

Exclusion Criteria:

* Pregnant or nursing females.
* Known hypersensitivity to fluoroquinolones or to any of the study ingredients.
* Use of any antibiotic within 72 hours of treatment.
* Any disease or condition that could interfere with the safety and efficacy evaluations of the study medications.
* Participation in an ophthalmic drug or device research study within 30 days prior to entry into the study.

Min Age: 1 Year | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 957 (Actual)
Dates: Start 2006-06; Primary Completion 2007-11 (Actual); Study Completion 2007-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Laura Trusso, Study Director — Bausch & Lomb Incorporated

REFERENCES:
- [Derived] DeCory HH, Sanfilippo CM, Proskin HM, Blondeau JM. Characterization of baseline polybacterial versus monobacterial infections in three randomized controlled bacterial conjunctivitis trials and microbial outcomes with besifloxacin ophthalmic suspension 0.6. PLoS One. 2020 Aug 25;15(8):e0237603. doi: 10.1371/journal.pone.0237603. eCollection 2020. PMID 32841261
- [Derived] Comstock TL, Paterno MR, Decory HH, Usner DW. Safety and tolerability of besifloxacin ophthalmic suspension 0.6% in the treatment of bacterial conjunctivitis: data from six clinical and phase I safety studies. Clin Drug Investig. 2010;30(10):675-85. doi: 10.2165/11536720-000000000-00000. PMID 20629472
- [Derived] Tepedino ME, Heller WH, Usner DW, Brunner LS, Morris TW, Haas W, Paterno MR, Comstock TL. Phase III efficacy and safety study of besifloxacin ophthalmic suspension 0.6% in the treatment of bacterial conjunctivitis. Curr Med Res Opin. 2009 May;25(5):1159-69. doi: 10.1185/03007990902837919. PMID 19323612

RESULTS

PARTICIPANT FLOW:
Recruitment Details: First subject enrolled 6/5/2006, last patient exited on 11/7/2007. This study was conducted at multiple sites in the US.
Pre-assignment Details: 957 Subjects with bacterial conjunctivitis were randomized to receive besifloxacin ophthalmic suspension or its vehicle, 11 subjects were discontinued due to failure to meet enrollment criteria or used disallowed medications.
Groups:
- ISV-403: Intraocular 0.6% ISV-403 ophthalmic suspension administered three times daily to affected eyes for 5 days.
- Vehicle: Vehicle of intraocular 0.6% ISV-403 ophthalmic suspension administered three times daily to affected eyes for 5 days.
Period: Overall Study
Arm/Group | ISV-403 | Vehicle
Started | 475 (As Randomized population - received at least one dose of study medication) | 482 (As Randomized Population - received at least one dose of study medication)
Completed | 444 | 430
Not Completed | 31 | 52
Not completed — Adverse Event | 4 | 5
Not completed — Lack of Efficacy | 3 | 14
Not completed — Lost to Follow-up | 10 | 9
Not completed — Withdrawal by Subject | 10 | 16
Not completed — Did not meet inclusion criteria | 4 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ISV-403 | Vehicle | Total
Number analyzed (Participants) | 475 | 482 | 957
Age, Customized [Number; unit: participants]
  <2 years | 21 | 20 | 41
  2 to 19 years | 196 | 196 | 392
  20 to 59 years | 212 | 226 | 438
  >=60 years | 46 | 40 | 86
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 302 | 300 | 602
  Male | 173 | 182 | 355
Race/Ethnicity, Customized [Number; unit: Participants]
  Caucasian | 312 | 312 | 624
  Asian | 10 | 7 | 17
  Black or African American | 44 | 46 | 90
  Other | 109 | 117 | 226
Region of Enrollment [Number; unit: participants]
  United States | 475 | 482 | 957

OUTCOME MEASURES:

1. Primary Outcome: Clinical Resolution of Baseline Bacterial Conjunctivitis
Description: The absence (grade 0 on the ordinal scale) of ocular discharge and bulbar conjunctival injection
Time Frame: Day 5 +/- 1 day
Population: Modified intent to treat population, culture confirmed, as randomized
Measure: Number; unit: Participants
Arm/Group | ISV-403 | Vehicle
Number analyzed (Participants) | 199 | 191
Participants | 90 | 63

2. Primary Outcome: Microbial Eradication of Baseline Bacterial Infection
Description: Absence (grade 0 on the ordinal scale) of all ocular bacterial species that were present at or above the threshold value for that species from the Cagle list at baseline.
Time Frame: Day 5 +/- 1 day
Population: Modified Intent to treat population, culture confirmed, as randomized.
Measure: Number; unit: Participants
Arm/Group | ISV-403 | Vehicle
Number analyzed (Participants) | 199 | 191
Participants | 182 | 114

3. Secondary Outcome: Clinical Resolution of Baseline Bacterial Conjunctivitis
Description: The absence (grade 0 on the ordinal scale) of ocular discharge and bulbar conjunctival injection
Time Frame: Day 8 or 9
Population: Modified intent to treat population, culture confirmed, as randomized
Measure: Number; unit: Participants
Arm/Group | ISV-403 | Vehicle
Number analyzed (Participants) | 199 | 191
Participants | 168 | 132

4. Secondary Outcome: Microbial Eradication of Baseline Bacterial Infection
Description: as for outcome 2
Time Frame: Day 8 or 9
Population: Modified intent to treat population, culture confirmed, as randomized.
Measure: Number; unit: Participants
Arm/Group | ISV-403 | Vehicle
Number analyzed (Participants) | 199 | 191
Participants | 176 | 137

ADVERSE EVENTS:
Time Frame: 8 days
Description: Treatment emergent ocular adverse events occured in < 5% of the patients
Arm/Group | ISV-403 | Vehicle
Serious Adverse Events (participants affected / at risk) | 1/442 | 1/432
Other Adverse Events (participants affected / at risk) | 0/741 | 0/760
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ISV-403 (N=442) | Vehicle (N=432)
Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Sponsor has 45 days to review materials and provide comments back to the investigator.